CLINICAL TRIAL: NCT04031170
Title: Filipino Family Health Initiative: The Incredible Years for Parents of School Age Children
Brief Title: Filipino Family Health Initiative
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Joyce Javier, Associate Professor, Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHLA-18-00066
Record Dates: First submitted 2018-12-12; First posted 2019-07-24 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Parenting; Family Relations; Education
Keywords: Filipino Families; Incredible Years

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Parents assigned to the intervention arm will receive the Incredible Years® School Age Basic & Advanced Parent Training Program. It consists of twelve (12) 2-hour classes led by Dean Coffey, a senior psychologist and certified peer coach in the Incredible Years Parent Training Series.
  Interventions: Behavioral: Incredible Years® School Age Basic Parent Training Program
- Control (Other): Parents assigned to the control arm will be emailed and mailed written parent education materials from the American Academy of Pediatrics called the Bright Futures handouts. The control group is offered the Incredible Years® School Age Basic & Advanced Parent Training Program after a 3-month wait list period.
  Interventions: Other: American Academy of Pediatrics, Bright Futures Handouts

INTERVENTIONS:
Behavioral: Incredible Years® School Age Basic Parent Training Program — The Incredible Years® School Age Basic Parent Training Program targets many of the proposed mechanisms and risk factors for internalizing distress in early childhood: harsh and unpredictable or critical parenting behaviors. Parents also learn cognitive strategies for themselves; such as self-praise, coping thoughts, how to challenge negative thoughts, and how to get support that they are encouraged to model for and teach their children. Finally, they learn how to be more positive and nurturing through academic, social and emotional coaching.
  Arms: Intervention
Other: American Academy of Pediatrics, Bright Futures Handouts — Written materials that include age-group specific tips on how parents can support their child's development and social and academic success.
  Other Names: Control
  Arms: Control

SUMMARY:
The overall objective of this research is to test the effectiveness of a parenting program on Filipino parents living in California. The sample will include 180 Filipino immigrant families, half of which will receive the Online Incredible Years® School Age Basic & Advanced Parent Training Program (intervention) and the other half will receive the American Academy of Pediatrics' Bright Futures handouts (control) and be placed on a 3-month waitlist for the IY parenting program.

DETAILED DESCRIPTION:
The overall objective of the proposed research is to test the effectiveness of a parenting program (Incredible Years® School Age Basic & Advanced Parent Training Program, IYP) on Filipino parents recruited from multiple community-based settings and its impact on trajectories of parenting practices, parenting stress, and child problem behavior.

Evidence-based parenting interventions provided in early childhood have proven to be effective in preventing the onset and escalation of child mental health disorders. IYP is one of the best-studied and most highly regarded parent training programs. As a result of pilot studies funded by a NIH K23 and a NCATS KL2 award, the investigators have identified IYP as a community-identified solution for preventing behavioral health disparities, demonstrated IYP efficacy in improving parenting practices and parenting stress in Filipino parents, and child problem behavior.

This population was chosen because: 1) Filipinos are the second largest immigrant population in the U.S. with the highest concentration living in Los Angeles; 2) Filipinos are exposed to multiple adversities, including immigration stress and relocation, loss of social status, and lower self-esteem due to discrimination, placing young children at risk for future behavioral and mental health problems; 3) U.S.-born Filipino youth exhibit higher rates of mental health problems than non-Hispanic whites and attain significantly lower levels of education than their foreign-born counterparts and other U.S.-born Asian American populations; and 4) Filipinos are less likely than non-Hispanic whites to participate in mental health and preventive care interventions.

The proposed study will be a randomized controlled trial involving 180 parents of children aged 8-12 years old. Parents will be randomly chosen to receive either a) an online 12 - week parenting intervention called the Incredible Years (intervention group) or b) AAP bright future handouts with general parenting advice (control group). The control group will be offered the Incredible Years after a 3-month wait list period.

Findings will contribute to the scientific literature on preventive and early intervention programs for children at high risk for future behavioral problems. The data will also provide important information to understand the processes underlying how IYP affects parenting practices and subsequent child problem behavior among Filipino families. The importance of this research rests on its potential to prevent behavioral health disparities in this understudied and high-risk population.

ELIGIBILITY:
NOTE: All parent participants in the study are 18 years or older. Youth participants are 8-12 years old. Since parents are the MAIN participants in this study (parents are randomized; children only fill out surveys), the age limits in this record are set for parents.

Inclusion Criteria:

* is 18 years or older
* identified as a parent of at least one Filipino or Half-Filipino child aged 8-12 years

Exclusion Criteria:

* if the parent plans to move out of California during the next 9 months
* parent does not speak English
* has a target child with a developmental disability (Global Developmental Delay, GDD), Pervasive Developmental Disorder (PDD), or another significant developmental condition)
* parent has completed Incredible Years school age program in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2018-07-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in parenting practices at 3 months in comparison to Baseline | Baseline and 3 months
  Parenting practices will be assessed using scores from the Parenting Practices Inventory (PPI). The PPI asks questions regarding parenting styles and behavior management techniques. Questions are rated on a scale ranging from never to always. A total score is not calculated.
Change in child behavioral problems at 3 months in comparison to Baseline | Baseline and 3 months
  Child problem behavior will be measured using scores from Child Behavior Checklist (CBCL). Parents describe their child's behavior within the past 6 months (from baseline and from 3 month time points). Questions are rated on a scale from 0 (not true) to 2 (very true or often true). The CBCL screens for the following behaviors: Aggressive Behavior, Anxious/Depressed, Attention Problems, Rule-Breaking Behavior, Somatic Complaints, Social Problems, Thought Problems, Withdrawn/Depressed. Results for each subscale are presented as a percentile and T-score, with scores above 97th percentile considered as "clinical range" based on the DSM-V.
Change in parenting practices at 6 months in comparison to Baseline and 3-month surveys | Baseline through 6 months
  Parenting practices will be assessed using scores from the Parenting Practices Inventory (PPI). The PPI asks questions regarding parenting styles and behavior management techniques. Questions are rated on a scale ranging from never to always. A total score is not calculated.
Change in child behavioral problems at 6 months in comparison to Baseline and 3-month surveys | Baseline through 6 months
  Child problem behavior will be measured using scores from Child Behavior Checklist (CBCL). Parents describe their child's behavior within the past 6 months. Questions are rated on a scale from 0 (not true) to 2 (very true or often true). The CBCL screens for the following behaviors: Aggressive Behavior, Anxious/Depressed, Attention Problems, Rule-Breaking Behavior, Somatic Complaints, Social Problems, Thought Problems, Withdrawn/Depressed. Results for each subscale are presented as a percentile and T-score, with scores above 97th percentile considered as "clinical range" based on the DSM-V.
Effectiveness of parenting workshop (Intervention group only): Incredible Years Parent Satisfaction Questionnaire | 3 months
  Consumer satisfaction will be assessed through the Incredible Years Parent Satisfaction Questionnaire. Consumer satisfaction will be assessed through the Incredible Years Parent Satisfaction Questionnaire. The questionnaire is rated on a 7-point scale ranging from unsatisfied extremely satisfied. A total score is not calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce R Javier, MD, MPH, MS, Principal Investigator — Children's Hospital Los Angeles, USC Keck School of Medicine
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be provided to the NIH National Institute of Mental Health Data Archives (NDA) repository. https://nda.nih.gov https://nda.nih.gov/nda/nimh-common-data-elements
  The NDA makes available human subjects data collected from hundreds of research projects across many scientific domains. NDA provides infrastructure for sharing research data, tools, methods, and analyses enabling collaborative science and discovery. De-identified human subjects data, harmonized to a common standard, are available to qualified researchers.

REFERENCES:
- [Derived] Javier JR, Aguiling W, Cunanan P, Sepulveda A, Coffey DM, Castro J, Palinkas LA, Kipke MD, Mack WJ. Short-term outcomes from a pilot randomized controlled trial evaluating a virtual culturally adapted parenting intervention among Filipino parents of school-age children. Cultur Divers Ethnic Minor Psychol. 2025 Jan;31(1):124-137. doi: 10.1037/cdp0000616. Epub 2023 Oct 19. PMID 37856386
- [Derived] Macam SR, Mack W, Palinkas L, Kipke M, Javier JR. Evaluating an Evidence-Based Parenting Intervention Among Filipino Parents: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2022 Feb 17;11(2):e21867. doi: 10.2196/21867. PMID 35175200